CLINICAL TRIAL: NCT04430829
Title: Comparison of Weight Bearing CT Arthrography With MRI for Detection of Knee Meniscal and Cartilage Lesions.
Brief Title: Diagnostic Value of Weight Bearing CT for Detecting Meniscal Tears
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Neil Segal, MD, MS, Director of Clinical Research, University of Kansas Medical Center
Other Study IDs: STUDY00145012
Record Dates: First submitted 2020-05-26; First posted 2020-06-12 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Meniscus Tear, Tibial
MeSH Terms: conditions — Tibial Meniscus Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Weight-Bearing CT arthrography — A 20ml mixture of 5ml 0.5% ropivacaine, 5ml preservative-free sterile saline, and 10ml of non-ionic iodinated contrast media (e.g. iohexol 240) will be instilled into the knee joint of each patient prior to WBCTa imaging of the knee (LineUp, CurveBeam, LLC).
Diagnostic Test: Knee MRI — MRI will be acquired (in-plane 0.25mm x 0.25mm, and 1.00mm slab thickness/separation and In-plane 0.25mm x 0.25mm, and 2.00mm slab thickness/separation)

SUMMARY:
This observational study will compare the clinical value of weight-bearing CT arthrography (WBCTa) with that for MRI in evaluating meniscal and cartilage lesions of the knee joint. The MRI Osteoarthritis Knee Score (MOAKS) and modified MOAKS for WBCTa will be used to compare findings between MRI and WBCTa of the knee while comparing with surgical measurements using the ICRS scoring system.

The study hypothesis is that meniscal and cartilage lesions may be missed by non-weight-bearing MRI, but detected by WBCTa.

DETAILED DESCRIPTION:
Study Objectives:

Aim 1 Establish the accuracy of WBCTa and MRI for diagnosing knee cartilage and meniscal lesions in both surgical and non-surgical participants.

Hypothesis 1: Pre-operative cartilage and meniscal scoring on WBCTa is more accurate than MRI, in comparison with arthroscopic assessment.

Aim 2 Establish the accuracy of WBCTa for detecting persistent and recurrent meniscal root and radial tears not detected by MRI 6 months after meniscal repair (defined by diastasis of the repair or meniscal extrusion ≥3mm).

Hypothesis 2: Six months following meniscal repair, WBCTa detects persistent and recurrent meniscal root and radial re-tears not detected by MRI.

Study Type and Design: This cross-sectional, observational study will compare WBCTa with MRI to evaluate rate of detection of meniscal and cartilage lesions. The inter-rater reliability of WBCTa readings also will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age with a knee MRI acquired in the previous 10 days to evaluate for suspected meniscal or cartilage pathology.
* Body mass index (BMI) ≤ 45 kg/m2
* Ability to stand with support without moving for at least 2 minutes.

Exclusion Criteria:

* End stage kidney disease
* Allergic to iodinated contrast material.
* Pregnancy
* Skin breakdown or rash at the knee joint which would prevent injection of the contrast.
* Any clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening which, in the opinion of the investigator, affects their ability to ambulate to a sufficient degree and could compromise patient safety or interfere with the assessment of the safety of the study injection.
* Superficial or deep infection in or around the index knee joint or allergy to iodinated contrast media.
* History of inflammatory arthritis, meniscectomy, or end-stage OA

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from orthopedic clinics as well as other musculoskeletal clinics that request knee MRI. Special efforts will be made to recruit the majority from orthopedic sports medicine clinical practices to include patients who are scheduled for arthroscopic meniscal repair of full-thickness radial tears of the posterior horn or body or root tears of the posterior horn after clinical MRI. There will be no exclusions based on sex or ethnic group.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
To determine the agreement between weight-bearing CT arthrography (WBCTa) and MRI in evaluation of meniscal tears. | Baseline
  Pre-operative cartilage lesion scoring of meniscal lesions on WBCTa (modified MOAKS score) and MRI (modified MOAKS score) will be compared with arthroscopic visual MOAKS scoring of meniscal lesions.

SECONDARY OUTCOMES:
To determine the agreement between weight-bearing CT arthrography and MRI in evaluation of cartilage lesions. | Baseline
  Musculoskeletal radiologists, each with greater than 10 years of experience will assess the morphology of the medial and lateral tibiofemoral cartilage on MRI and WBCTa using the MOAKS scoring system. Area of cartilage damage per subregion will be graded according to the MOAKS classification from 0-3: 0= no cartilage damage, 1=cartilage damage involving <10% of the subregion area, 2= cartilage damage involving 10%-75% of the subregion area and 3=cartilage damage involving >75% of the subregion area. The scores will be compared by dichotomizing into lesion present/absent (primary) and also compared using the full ranges of ordinal scores.
To determine the extent to which WBCTa identifies meniscal re-tears or failed repairs 6 months following meniscal root or radial tear surgical repairs | 6 months
  Participants who undergo a meniscal repair for radial meniscal tears and posterior root tears will undergo 6-month post-operative MRI and WBCTa and each of these 2 imaging modalities will be assessed for visualization of the presence or absence of a meniscal tear..

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, MS, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided